CLINICAL TRIAL: NCT00424931
Title: A Phase II Randomized, Double-blind, Double-dummy, Placebo and Comparator-controlled, Parallel Group, Multi-Center Study to Investigate the Safety and Efficacy of a Single Dose of JNJ-17216498 Administered to Subjects With Narcolepsy.
Brief Title: A Safety and Effectiveness Study of a Single Dose of JNJ-17216498 in Patients With Narcolepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alza Corporation, DE, USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR013390; C-2006-028
Record Dates: First submitted 2007-01-19; First posted 2007-01-22 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2014-05

CONDITIONS: Narcolepsy
Keywords: narcolepsy; sleepiness
MeSH Terms: conditions — Narcolepsy; Sleepiness | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- 001 (Experimental): JNJ-17216498 10mg one time
  Interventions: Drug: JNJ-17216498
- 002 (Experimental): JNJ-17216498 50mg one time
  Interventions: Drug: JNJ-17216498
- 003 (Active Comparator): Modafinil 200 mg X 2
  Interventions: Drug: Modafinil

INTERVENTIONS:
Drug: JNJ-17216498 — 50mg one time
  Arms: 002
Drug: JNJ-17216498 — 10mg one time
  Arms: 001
Drug: Modafinil — 200 mg X 2
  Arms: 003

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of JNJ-17216498 compared to modafinil and placebo in patients with narcolepsy, with and without cataplexy.

DETAILED DESCRIPTION:
This study with a new, experimental drug is being done to assess safety and tolerability, and to explore effectiveness in the treatment of narcolepsy. Approximately 64 adult patients with narcolepsy with or without cataplexy will be recruited for the study. Patients who meet study criteria will need to stop taking their current narcolepsy and/ or other medication for at least 14 days before checking into the site for 3 nights. They will be randomly assigned to one of 4 treatment arms; each patient has an equal chance of receiving placebo, 10 mg JNJ-17216498, 50 mg JNJ-17216498 or 400 mg modafinil. Placebo has no active drug. Modafinil is a drug currently approved to treat narcolepsy. Patients will take the medication on only one day and will receive study medication in a blinded fashion, i.e. the patient, the doctor and the study sponsor will not know what group the patient is in until all patients complete the study. The investigator and the sponsor will monitor the study for the occurrence of possible side effects. In addition to a screening visit and the three nights at the site, there will be a follow-up visit 7-10 days after the day the study drug is taken. After the follow-up visit, patients may resume their previous narcolepsy medications. Medical history, physical examination, vision tests, blood pressure, heart rate, temperature, and ECGs will be checked periodically. Blood samples will be taken for standard safety laboratory tests as well as for the measurement of the drug blood level. The Maintenance of Wakefulness Test will be done to assess the patient's ability to resist falling asleep while reclining in a dark, quiet room; this will involve completing 7 sessions before dosing and 10 sessions after dosing. Patients will have two polysomnograms, a test of brain, muscle and eye activity during sleep, obtained by recording brain waves and other activities such as muscle and eye movement. Polysomnograms will be obtained overnight, once before and once after dosing. Patients will also complete brief questionnaires about their sleepiness and the status of their narcolepsy throughout the study. Patients will receive capsules containing either 10 mg JNJ-17216498, 50 mg JNJ-17216498, 400 mg modafinil and/or placebo on one day. Seven capsules will be taken orally in the morning and two capsules will be taken orally in the afternoon. Placebo contains no active drug. Modafinil is a drug currently approved to treat narcolepsy.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of narcolepsy within the past 5 years
* good general health
* no history or presence of drug or alcohol abuse

Exclusion Criteria:

* current use of prescription or over the counter medications including asprin or herbal supplements with the exception of acetaminophen (Tylenol)
* use of fluoxetine (Prozac) in the past 6 weeks
* use of Xyrem in the past 4 weeks
* use of tobacco products in the past 3 months
* caffeine consumption that is more than 5 cups of tea, or 3 cups of coffee or 8 cans of soda per day

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2007-01; Primary Completion 2007-11 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Explore the effectiveness of JNJ-17216498 in patients with narcolepsy as determined by the Maintenance of Wakefulness Test done throughout the study. | ·To explore efficacy of JNJ-17216498 in patients with narcolepsy with or without cataplexy up through 48 hours after dosing.

SECONDARY OUTCOMES:
Explore the safety and tolerability of JNJ-17216498 in patients with narcolepsy by assessing adverse events, vital signs, laboratory results, vision tests, physical exam and ECGs. | To explore the safety and tolerability of JNJ-17216498 in patients with narcolepsy with or without cataplexy throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — ALZA
Locations (16):
- United States (16):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - San Diego, California
  - Stanford, California
  - Spring Hill, Florida
  - St. Petersburg, Florida
  - Macon, Georgia
  - Danville, Indiana
  - Fort Wayne, Indiana
  - Amherst, New York
  - Cincinnati, Ohio
  - Toledo, Ohio
  - Columbia, South Carolina
  - Houston, Texas
  - Spokane, Washington